CLINICAL TRIAL: NCT02276963
Title: Phase I, Single-Center, Open Label Trial of Ublituximab + Glucocorticoids for the Treatment of Acute Optic Neuritis and/or Transverse Myelitis in Neuromyelitis Optica (NMO) and Neuromyelitis Optica Spectrum Disorder (NMOSD)
Brief Title: Ublituximab for Acute Neuromyelitis Optica (NMO) Relapses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00052958
Record Dates: First submitted 2014-10-21; First posted 2014-10-28 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Neuromyelitis Optica; Neuromyelitis Optica Spectrum Disorder
Keywords: Transverse myelitis, optic neuritis, neuromyelitis optica
MeSH Terms: conditions — Neuromyelitis Optica; Myelitis, Transverse; Optic Neuritis | interventions — ublituximab; LFB-R603

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ublituximab Plus Glucocorticoids (Experimental): Ublituximab 450 mg intravenously once on day 1, plus glucocorticoids 1000 mg intravenously daily on days 1-5
  Interventions: Drug: Ublituximab

INTERVENTIONS:
Drug: Ublituximab — Monoclonal antibody that specifically binds to the trans-membrane antigen CD20, which induces immune response that causes lysis of B cells.
  Other Names: LFB-R603

SUMMARY:
Ublituximab (also known as LFB-R603) is a monoclonal antibody that specifically binds to the trans-membrane antigen CD20. The binding induces immune response that causes lysis of B cells.

The rationale for using ublituximab in neuromyelitis optica (NMO) and neuromyelitis optica spectrum disorder (NMOSD) is based on the known roles of B cells, antibody production and plasma cells in the pathophysiology of NMO. NMO is characterized by the presence of an anti-Aquaporin-4 (AQP4) antibody, which can only be produced by differentiation of B cells to plasma cells. Because these anti-AQP4 antibodies may be pathogenic, B cells recognizing AQP4 may be directly involved in the disease process as well. B cells also play a role as potent antigen presenting cells in NMO. The strongest evidence of the importance of B cells in NMO comes from studies of B cell depletion, most commonly with anti-CD20 monoclonal antibody, rituximab (Rituxan®).

Rituximab has been shown in five retrospective and two prospective studies to be effective in reducing NMO relapses up to 90% and achieving remission in up to 80% of patients solely by its action on CD20+ B cells, despite no change in plasma cell population and anti-AQP4 antibody titers. These human trials strongly suggest a critical role for B cells in the pathophysiology of human disease. While typically used in the prevention of disease, B-cell depletion may be beneficial in the treatment of an acute relapse as well. Emerging evidence indicates that peripheral B cells are activated during a relapse and plasmablast production of anti-AQP4 antibodies spikes. B cells are also found within acute lesions of the spinal cord and optic nerve suggesting roles both in the blood and in the central nervous system during a relapse.

DETAILED DESCRIPTION:
The overall objective is to assess the safety of ublituximab as add-on therapy to steroids for treatment of acute optic neuritis and/or transverse myelitis in NMO and NMOSD.

Primary Objective To assess safety of acute B cell depletion in NMO subjects with acute relapse of optic neuritis or transverse myelitis who are treated with ublituximab + glucocorticoids beginning on dose administration and ending with recovery of B cells.

Secondary Objectives

* To determine the B cell depletion pharmacokinetics of ublituximab in the NMO patients population with monthly B cell counts for up to 9 months.
* To determine the frequency of adverse events with ublituximab in this patient population.

Trial Design Given the severity and the consequences of relapse in NMO, placebo treatment without steroid treatment is unethical and use of an active treatment is considered mandatory. The potential of currently utilized drugs and techniques to reduce the inflammation in NMO has been established primarily through expert consensus and small open label and retrospective studies.

This is a Phase 1 open-label, standard-of-care, single treatment arm, unblinded, single center interventional trial in NMO/NMOSD patients in which experimental subjects will receive one (1) infusion of 450 mg of intravenous ublituximab at the onset of an NMO exacerbation in addition to standard of care treatment with daily intravenous glucocorticoid at 1000 mg for five days.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent.
2. 18-100 years of age.
3. New acute optic neuritis and/or transverse myelitis. A clinical event is defined as an episode of inflammation in the spinal cord and/or optic nerve leading to neurologic deficits on physical exam not attributable to another disease process.
4. Confirmed or highly suspected diagnosis of NMO according to the 2006 revisions of the Wingerchuk diagnostic criteria for NMO (Wingerchuk, 2006), or AQP4 positive NMOSD.
5. The B cell count must be normal (5-20% of total lymphocytes) in subjects who have not received another B cell depleting therapy in the past year. For those on B cell depleting therapy within the past year, a B cell count of at least 0.5% is necessary.
6. A female subject is eligible to enter the trial if she is:

   * Not pregnant or nursing;
   * Of non-childbearing potential OR of child-bearing potential
7. Subject has a negative serum pregnancy test at screening and agrees to one of the following:

   * Complete abstinence from intercourse for the period from consent into the trial until 6 months after the last dose of investigational product; or,
   * Consistent and correct use of one of the following acceptable methods of birth control for the period from consent into the trial until 6 months after the last dose of investigational product:

     * Oral contraceptives
     * Injectable progesterone
     * Levonorgestrel implants
     * Estrogenic vaginal ring
     * Percutaneous contraceptive patches
     * Intrauterine device (IUD) or intrauterine system (IUS)
     * Male partner sterilization
     * Double barrier method

Exclusion Criteria:

1. Current evidence or known history of clinically significant infection including:

   * Chronic or ongoing active infectious disease
   * Previous serious opportunistic or atypical infections.
   * Hepatitis B
   * Tuberculosis (TB)
   * HIV
2. History of clinically significant central nervous system (CNS) trauma (e.g. spinal cord compression).
3. Past or current history of medically significant adverse effects from:

   * Corticosteroids
   * Diphenhydramine
   * Murine or mouse/human chimeric antibodies
4. Past or current malignancy, except for

   * Cervical carcinoma Stage 1B or less
   * Non-invasive basal cell and squamous cell skin carcinoma
   * Cancer diagnoses with a duration of complete response (remission) >5 years A history of hematologic malignancy excludes a subject from participation, regardless of response.
5. Significant concurrent, uncontrolled medical condition including, but not limited to, cardiac, renal, hepatic, hematological, gastrointestinal, endocrine, immunodeficiency syndrome, pulmonary, cerebral, psychiatric, or neurological disease which could affect the subject's safety, impair the subject's reliable participation in the trial, impair the evaluation of endpoints, or necessitate the use of medication not allowed by the protocol, as determined by the PI of the trial.
6. Use of an investigational drug or other experimental therapy for a condition other than NMO within 4 weeks, 5 pharmacokinetic half lives or duration of biological effect (whichever is longer) prior to screening.
7. Current participation in any other interventional clinical trial. Participation in non-interventional trial requires approval of the protocol by investigator.
8. Subjects who are concurrently receiving any other investigational agents, or have participated in an interventional clinical trial within the last 21 days, or subjects who have been vaccinated with a live vaccine < 2 months prior to trial inclusion.
9. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ublituximab breastfeeding should be discontinued if the mother is treated with ublituximab.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2019-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Levy, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single center, phase I open label study of ublituximab in NMOSD patients with acute relapses. Patients aged 18-65 who presented to the Johns Hopkins Hospital between January and September 2016 with new neurologic symptoms were eligible for enrollment if they demonstrated a new contrast-enhancing lesion on MRI.
Pre-assignment Details: There were no pre-assignment events.
Period: Overall Study
Arm/Group | Ublituximab Plus Glucocorticoids
Started | 6
Completed | 3
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: 1 patient withdrew from the study prior to exposure to drug. 5 subjects were exposed to the drug. 3 patients completed the study with monthly blood tests and 90 day follow up.
Arm/Group | Ublituximab Plus Glucocorticoids
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
AQP4 IgG serostatus [Count of Participants; unit: Participants] — Patient with neuromyelitis optica spectrum disorder are stratified by presence of a serological antibody (IgG) to Aquaporin-4 (AQP4), seropositive and seronegative.
  Participants
    AQP4 IgG seropositive | 5
    AQP4 IgG seronegative | 0
Duration of disease [Mean (Standard Deviation); unit: years] | 12.2 (4.5)
Number of previous relapses [Mean (Standard Deviation); unit: relapses] | 4.8 (1.3)
Background immunotherapy [Count of Participants; unit: Participants] — Patients diagnosed with neuromyelitis optica spectrum disorder are recommended off label immunotherapy to try to prevent relapses. Although some of the patients were on such immunotherapies, they failed to prevent relapses. However, they may have an impact on the severity or recovery process.
  Participants
    None | 2
    Mycophenolate mofetil | 2
    Rituximab | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Neurological Disability - Expanded Disability Scale Score
Description: The Kurtzke Expanded Disability Status Scale (EDSS) was developed to measure the disability status of subjects with demyelinating disease. It allows an objective quantification of the level of functioning that could be widely and reproducibly used by researchers and health care providers. The EDSS provides a total score on a scale that ranges from 0 to 10 where 0 is normal and 10 is deceased. Increasing disability is reflected in an increasing EDSS score.
Time Frame: On admission to the hospital on day 1, on discharge 5-21 days later and on follow up at 90 days
Population: 5 subjects had EDSS measurements at the first three time points: baseline, admission and discharge. 3 subjects had EDSS scores with an additional EDSS measurement at 90-day follow up.
Measure: Median (Inter-Quartile Range); unit: EDSS unit score
Arm/Group | Ublituximab Plus Glucocorticoids
Number analyzed (Participants) | 5
EDSS unit score
  Baseline | 4.0 [2.25 to 5.5]
  Admission | 6.5 [5.25 to 7.5]
  Discharge | 6.5 [4.75 to 7.5]
  90-day follow up: number analyzed (Participants) | 3
  90-day follow up | 4.0 [2.0 to 8.0]

ADVERSE EVENTS:
Time Frame: 90 days
Description: Definition: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Ublituximab Plus Glucocorticoids
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 3/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ublituximab Plus Glucocorticoids (N=5)
Headache/body ache (Musculoskeletal and connective tissue disorders) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT02276963/Prot_SAP_000.pdf
  • Informed Consent Form (2015-09-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT02276963/ICF_001.pdf